CLINICAL TRIAL: NCT05572606
Title: Development and Delivery of a Novel Hypnotherapy Protocol for Treatment of Symptomatic Bloating
Brief Title: Treatment of Symptomatic Bloating Using a Novel Hypnotherapy Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Xiao Jing (Iris) Wang, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-005844
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Bloating
Keywords: Hypnotherapy
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypnotherapy for bloating symptoms (Experimental): Subjects experiencing bloating symptoms will receive hypnotherapy delivered electronically
  Interventions: Behavioral: Hypnotherapy

INTERVENTIONS:
Behavioral: Hypnotherapy — Seven pre-recorded hypnotherapy sessions delivered over the course of twelve weeks via the patient's own electronic device such as a smartphone, tablet, or laptop. The length of the audio-recorded treatment sessions is expected to be approximately 40 minutes on average.

SUMMARY:
The purpose of this research is to evaluate if hypnotherapy delivered electronically will help with bloating symptoms.

DETAILED DESCRIPTION:
This study consists of seven pre-recorded hypnotherapy sessions that will be digitally delivered to patients on their own electronic devices via an existing digital platform provided by metaMe Health. metaMe Health is a company specialized in the delivery of digital hypnotherapy protocols. The sessions will be delivered to patients over twelve weeks in accordance with current gut-direct hypnotherapy practice. The patients must agree to have their consent and content delivered electronically and provide periodic outcomes by completing electronic symptom questionnaires. The whole study will last for 24 weeks: the initial 12-week treatment period and then an additional 12-week follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Patients who meet Rome IV criteria for functional abdominal bloating/distension.
* Patients who meet criteria for other Rome IV Disorder of Gut Brain Interaction diagnoses (including but not limited to irritable bowel syndrome, functional constipation, or functional dyspepsia) may be included if bloating is their predominant symptom.
* Patients will be proficient in English language for comprehension of content.
* Patients will have reliable access to digital delivery systems for content and questionnaire access via smartphone over the course of the study and follow up period.

Exclusion criteria:

* Patients with known prior diagnosis of small intestinal bacterial overgrowth (SIBO), gastroparesis, rumination syndrome, chronic intestinal pseudo-obstruction, advanced connective tissue diseases (e.g., scleroderma), and uncontrolled inflammatory bowel disease (IBD) will be excluded.
* Patients with known disaccharide intolerances may be included if dietary restrictions are maintained during the duration of the study.
* Patients who have a history of cognitive delay, traumatic brain injury with residual deficits, history of cerebral vascular accident with residual deficiencies in cognition, dementia, shall be excluded.
* Patients with significant psychiatric illness with component of psychosis (schizophrenia, bipolar disorder), as well as severe untreated major depressive disorder with suicidal ideation will be excluded.
* Patients with substance abuse disorders and drug addiction will be excluded.
* Patients who are unlikely to comply or unlikely to benefit from psychotherapy-based interventions may be excluded at the direction of medical screening provider or principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in abdominal bloating severity | Baseline, 6 weeks, 12 weeks, and 3 months
  Measured on a 0-100 scale using the bloating severity question of the the validated Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS)

SECONDARY OUTCOMES:
Bloating symptoms | Baseline, 6 weeks, 12 weeks, and 3 months
  Assessed using the well validated upper GI symptom Severity Index (PAGI-SYM)
Change in perception of GI symptoms | Baseline, 6 weeks, 12 weeks, and 3 months
  Measured using the self-reported Visceral Sensitivity Index (VSI)
Change in quality of life | Baseline, 6 weeks, 12 weeks, and 3 months
  Assessed via the self-reported EuroQol-5D-5L (EQ-5D-5L) to evaluate mobility, self-care, usual activity, pain/discomfort, and anxiety/depression
Health care utilization | Baseline, 12 weeks, and 3 months
  Assessing the number of outpatient visits, portal messages, and procedures generated in three months

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Jing (Iris) Wang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials